CLINICAL TRIAL: NCT00152672
Title: Treatment of Sleep Apnea Syndrome With nCPAP Versus Oral Appliance: a Multicentre Prospective Randomized Crossover Trial
Brief Title: Treatment of Sleep Apnea Syndrome With nCPAP Versus Oral Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 04-10
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-02

CONDITIONS: Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

INTERVENTIONS:
Device: nCPAP vs oral appliance

SUMMARY:
This prospective randomized cross over study aims to compare nCPAP with mandibular advancement device for the treatment of sleep apnea syndrome.The effectiveness of nCPAP and oral appliance on apnea-hypopnea index, daytime sleepiness and quality of life will be compared in 60 patients.

ELIGIBILITY:
Inclusion Criteria:

18 to 70 years old BMI < 35 kg/m2 Apnea-hypopnea index between 10 and 60 events/h Complaint of snoring and sleepiness Dental status adequate for treatment with oral appliance informed consent

Exclusion Criteria:

psychiatric disease professional driver other cause of sleepiness

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Gagnadoux, Principal Investigator — UH Angers
Locations (1):
- CHU, Angers, France